CLINICAL TRIAL: NCT02298231
Title: Improving Balance in TBI Using a Low-Cost Customized Virtual Reality Rehabilitation Tool
Brief Title: Improving Balance in TBI Using Virtual Reality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: Fort Belvoir Community Hospital (U.S. Federal Agency); University of Southern California (Other); VA Office of Research and Development (U.S. Federal Agency); Kessler Institute for Rehabilitation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-831-14
Record Dates: First submitted 2014-11-05; First posted 2014-11-21 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Balance; TBI; Veterans; Virtual Reality
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Group 1 (Experimental): Standard of Care Balance (SCB) Treatment
  Interventions: Other: Standard of Care Balance Intervention
- Group 2 (Experimental): Mystic Isle (MI) Balance Training
  Interventions: Other: Mystic Isle Balance Intervention
- Group 3 (Experimental): Mystic Isle (MI) Dual Task Training
  Interventions: Other: Mystic Isle Balance Intervention with Dual Task

INTERVENTIONS:
Other: Standard of Care Balance Intervention — Standard balance therapy as performed by a physical therapist
  Arms: Group 1
Other: Mystic Isle Balance Intervention — Balance therapy using virtual reality
  Arms: Group 2
Other: Mystic Isle Balance Intervention with Dual Task — Balance therapy using virtual reality and performing cognitive tasks
  Arms: Group 3

SUMMARY:
This research study evaluates the effectiveness of a low-cost Virtual Reality-based (VR) training system in providing a customized balance treatment in a skilled clinical setting. Participants will be assigned to one of three treatment groups.

DETAILED DESCRIPTION:
Traumatic Brain injury (TBI) is a major health concern for the U.S. military and civilian populations, resulting in more than 5.3 million people who require rehabilitation and assistance for the short and long-term consequences of TBI. TBI impairs the integration and organization of the visual, auditory and somatosensory inputs that permit body position awareness, in relation to self and the environment. Even minor impairments in any of these systems can cause balance dysfunction (BDF), which is one of the most disabling aspects of TBI. BDF affects over 65% of all individuals with TBI. When cognitive deficits are present, BDF may become more pronounced, particularly when attempting to engage in more than one task at a time (i.e., dual task). Treating BDF in patients with TBI can be challenging, as traditional treatments do not consistently replicate everyday life environments. Virtual reality (VR) interventions enable clinicians to systematically deliver and control dynamic, interactive, multisensory stimuli. The proposed study will implement and evaluate a novel, low-cost, VR rehabilitation tool (Mystic Isle; MI) targeting somatosensory, vestibular, and vision systems through a double-blind RCT. Given the importance of dual-task skills for real-world functioning, the investigators will also evaluate the relative effectiveness of dual task (balance and cognitive) VR training to improve balance.

Preliminary case, feasibility and efficacy studies have been conducted using MI with rehabilitation populations. Findings demonstrate that customized VR using full-body movement tracking is motivating, feasible for balance training in neurorehabilitation populations, and results in improved balance and motor action planning. The proposed study will directly evaluate the effectiveness of a low-cost, interactive, multisensory, VR training using MI to improve balance and global functioning. The investigators will evaluate the relative effectiveness of dual task (balance and cognitive) VR training to improve balance, the long-term effectiveness of such training, and the utility of a balance maintenance program for facilitating longer-term treatment effects.

A total of 180 participants (Service Members, Veterans, civilians) with mild to severe TBI and documented balance impairments will be randomly assigned into one of three balance treatment groups: 1) Standard of care (control condition); 2) MI; 3) MI dual task (balance plus cognitive). All groups will undergo 2 treatment sessions/week x 6 weeks (i.e. 12 sessions). Following completion of the treatment protocol, participants in the MI training group will be randomly assigned to a maintenance training group (2 sessions/month x 4 months) or a non-maintenance group. All participants will undergo baseline, immediate (6 weeks), and long-term (4 months) follow-up assessments of: 1) static and dynamic balance and 2) community integration, self-efficacy, quality of life, and cognitive function. This design will allow us to assess the efficacy of MI as a customizable balance treatment in TBI, and to evaluate the impact of this remediation program on overall functioning.

The following hypotheses are proposed: 1) Participants completing both MI training conditions will exhibit significantly improved balance relative to the control group; 2) Participants completing both MI training conditions will demonstrate significantly greater improvements in global functioning relative to the control group; 3) Participants receiving the MI dual task training (balance and cognitive) will exhibit significantly greater improvements in balance relative to those in the single task MI training; 4) Participants completing both MI training conditions will sustain treatment gains for up to 4 months following treatment relative to baseline performance; the control group will maintain or decrease balance between follow-up sessions; and 5) Participants receiving maintenance training will maintain better balance over the 4 month follow-up period compared to the non-maintenance group.

The proposed study is poised to make an important contribution to enhancing balance function in service members and civilians with TBI, thereby promoting recovery of physical and social functioning and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with a mild to severe Traumatic Brain Injury (TBI). My TBI severity will be categorized by research study staff based on length of loss of consciousness (LOC), alteration of consciousness/mental state (AOC) or post-traumatic amnesia (PTA).
* Must be out of PTA, as indicated by O-log score of > 24 on 2 consecutive days as determined by study staff.
* Be at least 3 months post injury.
* Speak English.
* As determined by study personnel, have at least 20/60 acuity in worst eye according to the Snellen Eye Exam.
* As determined by study personnel, receive an acceptable score on the Token Test.
* Balance dysfunction as determined by impairment on standing balance measures (Sensory Organization Test)
* Be able and willing to comply with study procedures, including follow-up requirements.
* Be willing and able to give informed consent

Exclusion Criteria:

* Have an unstable or uncontrolled seizure disorder.
* Have a diagnosis of excessive fluid surrounding my brain.
* Have severe cardiac disease (e.g. heart attack or heart failure).
* Have uncontrolled or unstable orthostatic hypotension (blood pressure drops suddenly when one stands, causing one to feel light headed or dizzy).
* Have had a lower limb injury in the past 90 days.
* Have any other injury that affects one's ability to balance.
* Have a pre-existing condition that significantly affects one's alignment or function of one's lower limb while standing.
* Be on any medication that may affect one's balance, strength, or muscle coordination (e.g. Botox, Baclofen).
* Have significant neurological history (e.g.epilepsy that began before TBI, multiple sclerosis) other than TBI.
* Have significant psychiatric history (i.e. schizophrenia).
* Have a history of significant drug abuse.
* Have had physical or occupational therapy or treatment for balance disorder in the past 30 days.
* Have difficulty following or responding to commands that would limit study participation.
* Be currently enrolled in another research study that is likely to affect participation in this research study.
* Have any underlying medical conditions that would limit study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Balance Assessment | 4 months
  Physical tasks scored based on performance, e.g., 10 Meter walk, Balance Tasks and Computerized Sensory Organization Test

SECONDARY OUTCOMES:
Global Functioning evaluating the impact of the intervention on everyday life | 4 months
  Questionnaires
Neuropsychological Assessment examining changes in cognitive functioning | 4 months
  Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Nolan, PhD, Principal Investigator — Kessler Foundation; Denise Krch, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States